CLINICAL TRIAL: NCT00395720
Title: A Phase I Study Evaluating the Safety and Immunogenicity of a New TB Vaccine, MVA85A, in Healthy Volunteers Who Are Infected With HIV
Brief Title: The Safety and Immunogenicity of a TB Vaccine; MVA85A, in Healthy Volunteers Who Are Infected With HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB010
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Tuberculosis; HIV Infections
Keywords: TB; Tuberculosis; HIV; Vaccine; MVA85A; HIV Therapeutic Vaccine
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — MVA 85A; MVA Pfs25-IMX313 malaria vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Group 1 (10 volunteers): 5 x 10^7 pfu
  Interventions: Biological: MVA85A (TB vaccine); Biological: MVA 85A
- 2 (Active Comparator): Group 2 (10 volunteers): 1 x 10^8 pfu
  Interventions: Biological: MVA85A (TB vaccine); Biological: MVA 85A

INTERVENTIONS:
Biological: MVA85A (TB vaccine) — Intradermal vaccine
  Other Names: TB vaccine
Biological: MVA 85A — Intradermal vaccine
  Other Names: TB Vaccine; modified vaccinia virus Ankara

SUMMARY:
This study is designed to evaluate the safety of MVA85A in healthy volunteers in the UK who are infected with HIV. In phase I studies, a single vaccination with MVA85A, when administered at a dose of 5 x 10^7pfu intradermally, has been shown to be safe in both mycobacterially naïve individuals, those previously vaccinated with BCG and latently infected individuals. Additionally, 5 x 10^7 pfu MVA containing HIV antigens administered twice, 4 weeks apart, in HIV positive individuals, is safe. We will use 5 x 107 pfu MVA85A intradermally in this study. Subjects will be identified from HIV clinics in the Oxford Radcliffe Hospitals NHS Trust and also from Swindon and Marlborough NHS Trust and St. Mary's Hospital NHS Trust if our recruitment targets are not met.

DETAILED DESCRIPTION:
The need for new vaccine against tuberculosis Tuberculosis (TB) kills about three million people annually. It is estimated that one third of the world's population are latently infected with Mycobacterium tuberculosis (M.tb) (Dye, 1999). These latently infected individuals are at risk of reactivation of infection, should they become immunosuppressed. Worldwide, coinfection with HIV is the commonest cause of immunosuppression and increases the chances of reactivation from a 10% lifetime risk to a 10% annual risk (Corbett, 1996). The currently available vaccine, M. bovis BCG, is largely ineffective at protecting against adult pulmonary disease in endemic areas and it is widely agreed that a new more effective tuberculosis vaccine is a major global public health priority (Colditz, 1994). However, it may be unethical and impractical to test and deploy a vaccine strategy that does not include BCG, as BCG does confer worthwhile protection against TB meningitis and leprosy. An immunisation strategy that includes BCG is also attractive because the populations in which this vaccine candidate will need to be tested will already have been immunised with BCG. Given the high prevalence of infection with M.tb, a vaccine that could be administered to latently infected individuals and eradicate latent infection would have an enormous impact on the mortality and morbidity from TB. M.tb is an intracellular organism. CD4+ Th1-type cellular responses are essential for protection and there is increasing evidence from animal and human studies that CD8+ T cells also play a protective role (Flynn, 2001). However, it has generally been difficult to induce strong cellular immune responses in humans using subunit vaccines. DNA vaccines, recombinant viral vectors and protein/adjuvant combinations all induce both CD4+ and CD8+ T cells, however none of these antigen delivery systems induce high levels of antigen specific T cells, when used alone.

Heterologous prime-boost immunisation strategies involve giving two different vaccines, each encoding the same antigen, several weeks apart. Using a DNA prime-recombinant modified vaccinia virus Ankara (MVA) boost induces higher levels of antigen specific CD4+ and CD8+ T cells than using homologous boosting with the same vector in a number of different disease models (Schneider, 1998; McShane, 2001). Given the protective efficacy of BCG in childhood, ideally BCG would be the priming immunisation in such a prime-boost strategy. In order to do this, we have focused on antigen 85A as a candidate antigen. Antigen 85A is highly conserved amongst all mycobacterial species and is present in all strains of BCG. Antigen 85A is a major secreted antigen from M. tuberculosis which forms part of the antigen 85 complex (A, B and C). This complex constitutes a major portion of the secreted proteins of both M.tb and BCG. It is involved in fibronectin binding within the cell wall and has mycolyltransferase activity. Antigen 85A is immunodominant in murine and human studies and is protective in small animals (Huygen, 1996).

Recombinant modified vaccinia virus Ankara (rMVA). Many viruses have been investigated as potential recombinant vaccines. The successful worldwide eradication of smallpox via vaccination with live vaccinia virus highlighted vaccinia as a candidate for recombinant use. The recognition in recent years that non- replicating strains of poxvirus such as MVA and avipox vectors can be more immunogenic than traditional replicating vaccinia strains has enhanced the attractiveness of this approach. MVA (modified vaccinia virus Ankara) is a strain of vaccinia virus which has been passaged more than 570 times though avian cells, is replication incompetent in human cell lines and has a good safety record. It has been administered to more than 120,000 vaccinees as part of the smallpox eradication programme, with no adverse effects, despite the deliberate vaccination of high risk groups (Stickl, 1974; Mahnel, 1994). This safety in man is consistent with the avirulence of MVA in animal models. MVA has six major genomic deletions compared to the parental genome severely compromising its ability to replicate in mammalian cells (Meher, 1991). No replication has been documented in non- transformed mammalian cells. Viral replication is blocked late during infection of cells but importantly viral and recombinant protein synthesis is unimpaired even during this abortive infection. The viral genome has been proven to be stable through a large series of passages in chicken embryo fibroblasts. Replication-deficient recombinant MVA has been seen as an exceptionally safe viral vector. When tested in animal model studies recombinant MVAs have been shown to be avirulent, yet protectively immunogenic as vaccines against viral diseases and cancer. Recent studies in severely immuno-suppressed macaques have supported the view that MVA should be safe in immuno-compromised humans (Akira, 2001; Stittelaar, 2001). There is now safety data from a number of recombinant MVAs that are currently in Phase I/II trials in both the UK and Africa. Useful data on the safety and efficacy of various doses of a recombinant MVA vaccine comes from clinical trial data with a recombinant MVA expressing a number of CTL epitopes from Plasmodium falciparum pre-erythrocytic antigens fused to a complete pre-erythrocytic stage antigen, Thrombospondin Related Adhesion Protein (TRAP). To date MVA ME-TRAP has been administered to over 600 healthy volunteers (adults and children) in Oxford and Africa (The Gambia and Kenya) without any serious adverse events (Adrian Hill, unpublished, personal communication). Volunteers have received one to three doses of from 3 to 15 x 107 pfu per dose of intra-dermal vaccine at three-week intervals. All subjects have temporary local redness with typically a 5mm central red area with a paler pink surrounding area that ranges in size from about 1 -7cm in diameter and peaks at 48 hours post vaccination. At seven days post vaccination generally only the central red area remains. This fades over the next few weeks and is usually not apparent at 2 months after vaccination. The emerging safety profile of recombinant MVA vaccine is excellent and supported by data from clinical studies of three other MVA recombinants made in Oxford and currently in clinical studies using MVAs for HIV, HBV and melanoma. To date these vaccines have been administered to over 600 people with no serious adverse events (Hill; personal communication) 40 HIV positive individuals treated with highly active anti-retroviral therapy (HAART) have been vaccinated with at least 5 x 107 PFU MVA containing HIV antigens with no serious adverse events (Dorrell, unpublished data; Cosma et al 2003; Harrer et al, 2005). 7 HIV positive individuals have been vaccinated with MVA containing malaria antigens with no serious adverse events and no significant or sustained rise in viral load (Bejon at al, CID 2006, in press).

Recombinant MVA encoding antigen 85A MVA85A induces both a CD4+ and a CD8+ epitope when used to immunise mice. When mice are primed with BCG and then given MVA85A as a boost, the levels of CD4+ and CD8+ T cells induced are higher than with either BCG or MVA85A alone, and this regime is more protective than either vaccine alone (Goonetilleke et al, 2003). In the more sensitive guinea pig model, guinea pigs vaccinated with BCG, and then MVA85A, and then a second viral vector, fowlpox expressing antigen 85A, 6/6 guinea pigs are alive at the end of the experiment, compared with 2/6 guinea pigs vaccinated with BCG alone, and 0/6 control animals (Williams et al, 2005).

In rhesus macaques, this BCG prime-MVA85A and Fowlpox85A boost is more immunogenic than any of the vaccines alone, and is more protective than BCG alone (verrek et al, unpublished data).

Clinical studies using MVA85A MVA85A (at a dose of 5 x 107pfu) has been administered to 48 healthy volunteers in the UK, 21 healthy volunteers in The Gambia and 18 in South Africa, with no serious adverse events. We have designed our Phase I studies to allow for a vaccination of volunteer groups sequentially with a step-wise increase in mycobacterial exposure, in order to minimize the possibility of a Koch reaction. A Koch reaction describes the development of immunopathology in a person or animal with tuberculosis, when an exaggerated immune response to M.tb is stimulated. It was described in patients with TB disease when Koch performed his original studies employing mycobacteria as a type of therapeutic vaccination. It has now been demonstrated in the mouse model of therapeutic vaccination (Taylor, 2003). Available animal data suggest that these reactions do not occur in mice latently infected with M.tb, suggesting that such reactions may correlate with high bacterial load and that the Koch phenomenon may not pose a problem for vaccination of healthy albeit latently infected humans. We started these studies in healthy volunteers who were as mycobacterially naïve as possible. They were skin test negative and Elispot negative for PPD, ESAT 6 and CFP10, and had not had previously been vaccinated with BCG. We have now completed studies in the UK vaccinating volunteers previously vaccinated with BCG (McShane, Nature Med, 2004) and in The Gambia.

There are two ongoing studies in Oxford. The first is a phase I trial of the safety and immunogenicity of MVA85A in individuals who are latently infected with M.tb. We have now vaccinated all 12 volunteers with no serious adverse events. The second is a dose selection study evaluating the safety and immunogenicity of 2 different doses of MVA85A (1x10^8 and 1x10^7 pfu), in healthy adult volunteers who have previously been vaccinated with BCG. Here we have vaccinated 11 individuals with the higher dose (1x10^8) with no serious adverse events, the main side effect being a fever at 24-48 hours post-vaccination, which completely resolves over 24 hours. Results from the low dose arm will be collected over the next few months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Willingness to allow the investigators to discuss the volunteer's medical history with the volunteer's HIV lead physician (and GP, if appropriate)
* BCG vaccinated
* HIV antibody positive; diagnosed at least 6 months previously
* CD4 count >350; nadir CD4 not < 300
* HIV viral load not > 100,000 copies per millilitre
* Written informed consent

Exclusion Criteria:

* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or on urinalysis
* Any ARV therapy within the past 6 months
* Any AIDS defining illness
* CXR showing TB or evidence of other active infection
* Prior receipt of a recombinant MVA or Fowlpox vaccine
* Use of any investigational or non-registered drug, live vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune modifying drugs within six months of vaccination. (For corticosteroids, this will mean prednisolone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Presence of any underlying disease that compromises the diagnosis and evaluation of response to the vaccine (including evidence of cardiovascular disease, history of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ), history of insulin requiring diabetes mellitus, any ongoing chronic illness requiring ongoing specialist supervision (e.g., gastrointestinal), and chronic or active neurological disease)
* History of > 2 hospitalisations for invasive bacterial infections (pneumonia, meningitis)
* Suspected or known current drug and/or alcohol abuse (as defined by an alcohol intake of >42 units a week)
* Seropositive for hepatitis B surface antigen (HBsAg) and/ or hepatitis C (antibodies to HCV)
* Evidence of serious psychiatric condition
* Any other on-going chronic illness requiring hospital specialist supervision
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Pregnant/lactating female and any female who is willing or intends to become pregnant during the study
* Any history of anaphylaxis in reaction to vaccination
* PI assessment of lack of willingness to participate and comply with all requirements of the protocol, or identification of any factor felt to significantly increase the participant's risk of suffering an adverse outcome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Data on adverse events | 1 year

SECONDARY OUTCOMES:
Immune responses | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Dr, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Colditz GA, Brewer TF, Berkey CS, Wilson ME, Burdick E, Fineberg HV, Mosteller F. Efficacy of BCG vaccine in the prevention of tuberculosis. Meta-analysis of the published literature. JAMA. 1994 Mar 2;271(9):698-702. PMID 8309034
- [Background] McShane H, Brookes R, Gilbert SC, Hill AV. Enhanced immunogenicity of CD4(+) t-cell responses and protective efficacy of a DNA-modified vaccinia virus Ankara prime-boost vaccination regimen for murine tuberculosis. Infect Immun. 2001 Feb;69(2):681-6. doi: 10.1128/IAI.69.2.681-686.2001. PMID 11159955
- [Background] Huygen K, Content J, Denis O, Montgomery DL, Yawman AM, Deck RR, DeWitt CM, Orme IM, Baldwin S, D'Souza C, Drowart A, Lozes E, Vandenbussche P, Van Vooren JP, Liu MA, Ulmer JB. Immunogenicity and protective efficacy of a tuberculosis DNA vaccine. Nat Med. 1996 Aug;2(8):893-8. doi: 10.1038/nm0896-893. PMID 8705859
- [Background] Cosma A, Nagaraj R, Buhler S, Hinkula J, Busch DH, Sutter G, Goebel FD, Erfle V. Therapeutic vaccination with MVA-HIV-1 nef elicits Nef-specific T-helper cell responses in chronically HIV-1 infected individuals. Vaccine. 2003 Dec 8;22(1):21-9. doi: 10.1016/s0264-410x(03)00538-3. PMID 14604567
- [Background] Bejon P, Peshu N, Gilbert SC, Lowe BS, Molyneux CS, Forsdyke J, Lang T, Hill AV, Marsh K. Safety profile of the viral vectors of attenuated fowlpox strain FP9 and modified vaccinia virus Ankara recombinant for either of 2 preerythrocytic malaria antigens, ME-TRAP or the circumsporozoite protein, in children and adults in Kenya. Clin Infect Dis. 2006 Apr 15;42(8):1102-10. doi: 10.1086/501459. Epub 2006 Mar 14. PMID 16575727
- [Background] Goonetilleke NP, McShane H, Hannan CM, Anderson RJ, Brookes RH, Hill AV. Enhanced immunogenicity and protective efficacy against Mycobacterium tuberculosis of bacille Calmette-Guerin vaccine using mucosal administration and boosting with a recombinant modified vaccinia virus Ankara. J Immunol. 2003 Aug 1;171(3):1602-9. doi: 10.4049/jimmunol.171.3.1602. PMID 12874255
- [Background] McShane H, Pathan AA, Sander CR, Keating SM, Gilbert SC, Huygen K, Fletcher HA, Hill AV. Recombinant modified vaccinia virus Ankara expressing antigen 85A boosts BCG-primed and naturally acquired antimycobacterial immunity in humans. Nat Med. 2004 Nov;10(11):1240-4. doi: 10.1038/nm1128. Epub 2004 Oct 24. PMID 15502839